CLINICAL TRIAL: NCT07352514
Title: Use of PEA and Scutellaria in Synergy With Therapeutic Exercise in Chemotherapy-induced Peripheral Neuropathy (CIPN): a Clinical Trial
Status: Recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Other Study IDs: MFR032025
Record Dates: First submitted 2025-03-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN); Neuropathic Pain
Keywords: Chemotherapy-Induced Peripheral Neuropathy; Neuropathic Pain; Nutraceuticals; Palmitoylethanolamide; Scutellaria; Therapeutic Exercise; Cancer Patients; Pain Management; Neuropathy Treatment; Clinical Trial; Observational Case-Control Study
MeSH Terms: conditions — Neuralgia; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PEA + Scutellaria + Therapeutic Exercise: This group consists of patients who will receive a combination of palmitoylethanolamide (PEA) and Scutellaria along with a standardized therapeutic exercise regimen. The goal is to evaluate the synergistic effects of the nutraceuticals and exercise in reducing neuropathic pain and improving overall nerve health.
- Therapeutic Exercise Only: Patients in this group will participate in a standardized therapeutic exercise program without any additional nutraceutical intervention. This cohort will help determine the efficacy of therapeutic exercise alone in managing symptoms of chemotherapy-induced peripheral neuropathy (CIPN).
- PEA + Scutellaria Only: This group includes patients who will be treated with a combination of PEA and Scutellaria without participating in any structured exercise regimen. The aim is to assess the impact of the nutraceuticals alone on reducing neuropathic pain and improving nerve function.

SUMMARY:
This study aims to find out if taking specific dietary supplements (PEA and Scutellaria) along with therapeutic exercise can help reduce nerve pain and damage caused by chemotherapy. Many cancer patients experience nerve-related side effects from chemotherapy, which can significantly impact their quality of life. The study will observe patients who use these supplements and exercises to see if they can effectively manage and improve their nerve health and reduce pain.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a significant and common complication affecting 30-60% of cancer patients undergoing chemotherapy. CIPN results in damage to sensory, motor, autonomic, or cranial nerves, leading to debilitating neuropathic pain. This condition poses a substantial burden on healthcare resources and significantly impacts patients' quality of life. Effective management of neuropathic pain through pharmacological and rehabilitative treatments is crucial in both the acute and chronic phases.

The study aims to evaluate the efficacy of a combined treatment regimen involving nutraceuticals, specifically palmitoylethanolamide (PEA) and Scutellaria, along with therapeutic exercise, in patients suffering from post-chemotherapy peripheral neuropathy. The rationale behind this combination therapy is based on the anti-inflammatory and neuroprotective properties of PEA and Scutellaria, coupled with the beneficial effects of physical exercise on neuropathic pain and overall nerve health.

Study Design: This study is a clinical observational, prospective cohort study. Patients with CIPN due to chemotherapy will be enrolled and monitored over a period of time to observe the effects of the combined treatment on their neuropathic symptoms. The study is post-market and will not involve any investigational drugs. Patients will be divided into three treatment groups:

* Patients receiving PEA + Scutellaria + therapeutic exercise.
* Patients receiving only therapeutic exercise. . Patients receiving only PEA + Scutellaria.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Patients who have undergone chemotherapy treatment within the previous 6 months.
* Patients treated with PEA, Scutellaria, and standardized therapeutic exercise according to the EXCAP protocol from April 2025 to September 2025.
* Patients with a washout period from opioid-based analgesic therapy of at least 10 days or who are not receiving opioid-based analgesic therapy.
* Patients presenting with neuropathic pain (NRS ≥ 5).
* Patients able to provide written informed consent.

Exclusion Criteria:

* Patients younger than 18 years.
* Patients with hypersensitivity to PEA or any of the excipients listed in the Summary of Product Characteristics (SPC).
* Patients with diabetic pathology.
* Patients with severe hepatic impairment.
* Patients with severe disabilities that compromise the execution of therapeutic exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from adult patients (aged 18 years and older) attending oncology and neurology clinics at major hospitals in Palermo, Sicilia, Italia. These patients have undergone chemotherapy treatment within the last 6 months and are experiencing chemotherapy-induced peripheral neuropathy (CIPN). The source of the participants includes both the Oncology Department and the Pain Management Unit, ensuring a diverse and representative sample of the target population.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in Neuropathic Pain Intensity | Baseline; 30 days after intervention; 60 days after intervention
  The primary outcome measure is the reduction in the intensity of neuropathic pain as assessed by the Numerical Rating Scale (NRS) from baseline (day 0) to the first follow-up visit (day 30) and the second follow-up visit (day 60).This primary outcome measure evaluates the efficacy of the combined treatment regimen (PEA, Scutellaria, and therapeutic exercise) in reducing neuropathic pain in patients with chemotherapy-induced peripheral neuropathy.

SECONDARY OUTCOMES:
Reduction in Sensory Symptoms | Baseline; 30 days after intervention; 60 days after intervention
  Reduction in sensory symptoms such as dysesthesia and paresthesia, and improvement in thermal and proprioceptive sensitivity.These secondary outcome measures help evaluate the broader effects of the intervention, in addition to the primary focus on neuropathic pain reduction. If you need further assistance or additional details, feel free to let me know!
Improvement in Segmental Strength | Baseline; 30 days after intervention; 60 days after intervention
  Recovery of segmental strength as assessed by the Medical Research Council (MRC) Scale.
Adherence to Therapeutic Exercise | Baseline; 30 days after intervention; 60 days after intervention
  Evaluation of adherence to therapeutic exercise, measured by step count with pedometer, duration of exercise, and perceived exertion (RPE Scale).
Rate of Discontinuation | Up to 60 days (through study completion, up to 2 months)
  Assessment of the rate of discontinuation of the treatment regimen.These secondary outcome measures help evaluate the broader effects of the intervention, in addition to the primary focus on neuropathic pain reduction. If you need further assistance or additional details, feel free to let me know!

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. P. Giaccone, Palermo, Italia 90127, Palermo, Italia, Italy